CLINICAL TRIAL: NCT00457483
Title: A Cross-over Trial to Identify Patient Characteristics That Predict Blood Pressure Response to Antihypertensive Therapy in General Practice
Brief Title: Nijmegen Antihypertensive Management Improvement Study
Acronym: NAMIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: NAMIS
Record Dates: First submitted 2007-04-04; First posted 2007-04-06 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2011-04

CONDITIONS: Primary Hypertension
Keywords: hypertension; diuretic; angiotensin receptor blockers; prediction
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — Hydrochlorothiazide; Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: hydrochlorothiazide — 12.5 mg once-a-day
Drug: valsartan, 80 mg once-a-day — 80 mg once-a-day

SUMMARY:
High blood pressure is an important risk factor for diseases of heart and blood vessels like myocardial infarction and stroke. Many patients are not treated to target blood pressures, even though good blood pressure lowering drugs are available. Not all blood pressure drugs are equally effective in individual patients.

We hypothesize that individual patient characteristics can predict the best response on different blood pressure lowering drugs. In this study we will investigate whether a set of patient characteristics (anthropometric and laboratory) obtained before treatment may predict the blood pressure lowering response to representatives of two groups of drugs: those that inhibit renin-angiotensin system activity and those that decrease blood volume.

DETAILED DESCRIPTION:
Population-wide elimination of hypertension would reduce the incidence of all stroke, MI and heart failure with 30 to 50% and contribute to a reduction of between 25 to 50% of the total mortality related to these cardiovascular conditions. However, despite increasing numbers of antihypertensive medication prescriptions, hypertension control rates are still insufficient.

The current study will focus on improving the success rate of the initial treatment of hypertension. The individual response to antihypertensive drugs varies between individuals: many patients responding well to one drug respond poorly to another. We hypothesize this difference in response to depend on the presence of certain characteristics of patients, like waist circumference, age and gender.

The major objective of our study will be to identify patient characteristics that predict the efficacy of different classes of antihypertensive drugs. Despite pleas in international publications to tailor antihypertensive treatment on individual basis, until now patient characteristics are not taken into account in the medical treatment of hypertension. We will address our study objective by the use of a PRospective, Open label (medication not blind), Blinded End-point crossover design (PROBE) in which 100 general practice based, newly diagnosed hypertensive patients, aged 18 - 65 years will be included to be treated with a diuretic and an angiotensin receptor blocker (ARB). Each patient will be treated with standard doses of both medications consecutively. Treatment duration for each medication will be four weeks, with a four weeks washout period in between. The choice for a diuretic versus an ARB is based on the substantial difference in working mechanism representing the two major determinants of blood pressure: effect on intravascular volume (diuretic) or vascular tone (ARB). Blood pressures will be assessed with both 24 hour-monitoring and practice based standardized measurements.

Twenty-three different patient characteristics will be studied and were selected based on review of literature and pathophysiologic theory. These characteristics will be (1) simple anthropometric measures like body mass index and fat distribution, (2) demographic characteristics, such as gender or ethnicity or (3) disease characteristics such as baseline diastolic and systolic blood pressure, co-morbidity and blood plasma levels of easily measured bioactive compounds, like renin and B-type natriuretic peptide.

The primary outcome measure will be the difference in blood pressure response between both study drugs; secondary outcome measures will be the difference in the number of patients achieving target blood pressure and the number of adverse drug events.

We expect to find three to six significant patient characteristics that predict response to antihypertensive medication in terms of blood pressure reduction.

If our study indeed identifies relevant patient characteristics GPs will be able to initiate antihypertensive medical treatment more efficiently. We expect this will result in increased initial therapeutic success and reduction of the number of antihypertensive drugs needed. As a consequence we expect compliance and hypertension control rates to increase. These expectations will need to be confirmed in a general practice-based follow-up study on implementation in daily practice of the use of patient characteristics with compliance and hypertension control rates as outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years with newly diagnosed hypertension in general practice
* hypertension is defined as either > 140 mm Hg systolic or > 90 mm Hg diastolic on three separate days.

Exclusion Criteria:

* History of cardiovascular disease (transient ischemic attack (TIA), stroke, myocardial infarction (MI), peripheral arterial disease (PAD), atrial fibrillation (AF), angina pectoris (AP), Diabetes Mellitus)
* Unable to understand and/or speak Dutch
* Severe hypertension (> 200/120 mmHg)
* Irregular pulse
* Use of antihypertensive medication
* Contraindication to one of the trial drugs
* Serious suspicion on secondary hypertension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-08; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Blood pressure response as determined by Ambulatory Blood Pressure Monitoring | 4 week treatment period
Patient characteristics that predict this blood pressure response | 4 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Jaap Deinum, MD PhD, Principal Investigator — University Medical Center St Radboud Nijmegen; Carel Bakx, MD PhD, Principal Investigator — University Medical Center St Radboud Nijmegen
Locations (1):
- Nijmegen monitoring project coordinated from Nijmegen, Nijmegen, Netherlands

REFERENCES:
- [Derived] van der Wel MC, Biermans M, Akkermans R, Lenders JWM, van Weel C, Deinum J. Patient characteristics do not predict the individual response to antihypertensive medication: a cross-over trial. Fam Pract. 2018 Jan 16;35(1):67-73. doi: 10.1093/fampra/cmx075. PMID 28968870
- [Derived] van der Wel MC, Buunk IE, van Weel C, Thien TA, Bakx JC. A novel approach to office blood pressure measurement: 30-minute office blood pressure vs daytime ambulatory blood pressure. Ann Fam Med. 2011 Mar-Apr;9(2):128-35. doi: 10.1370/afm.1211. PMID 21403139